CLINICAL TRIAL: NCT04660773
Title: NARROW BAND UVB PHOTOTHERAPY VERSUS PREGABALIN IN TREATMENT OF REFRACTORY PRURITIS IN END STAGE RENAL DISEASE PATIENTS
Brief Title: PHOTOTHERAPY VERSUS PREGABALIN IN TREATMENT OF REFRACTORY UREAMIC PRURITIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, marwa eldeeb, lecturer of dermatology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0106476
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Refractory Uremic Pruritis
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NB UVB phototherapy (Active Comparator): (20 patients) will receive NB UVB phototherapy 3 sessions per week for 2 months.
  Interventions: Device: NB UVB phototherapy
- pregabalin (Active Comparator): 20 patients) will receive pregabalin oral therapy (50mg after each dialysis session) for 2 months.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Device: NB UVB phototherapy — ultraviolet phototherapy sessions
  Arms: NB UVB phototherapy
Drug: Pregabalin — oral medication
  Arms: pregabalin

SUMMARY:
Patients will be randomly assigned into 2 groups:

1. Group A: (20 patients) will receive NB UVB phototherapy 3 sessions per week for 2 months.
2. Group B: (20 patients) will receive pregabalin oral therapy (50mg after each dialysis session) for 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-60 years.
2. End stage renal disease (the last stage(stage 5) of chronic disease which means kidneys are only functioning at 10 to 15 percent of their normal capacity and dialysis or kidney transplant is necessary to stay alive).
3. Refractory uremic pruritis.

Exclusion Criteria:

1. Other causes of pruritis (Dermatological or systemic) e.g. atopic, cholestatic liver disease.
2. Photosensitivity.
3. Contraindication or allergy to pregabalin.
4. Patients on antipruritic drugs e.g. antihistamines, steroids, emollients, opioid agonists.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
5 D-itching scale | two month
  assessment of degree, duration, direction, disability and distribution of itching

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No